CLINICAL TRIAL: NCT02241018
Title: Mesenchymal Stem Cells Combined With CD25 Monoclonal Antibody and Calcineurin Inhibitors for Treatment of Steroid-resistant Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Brief Title: MSCs Combined With CD25 Monoclonal Antibody and Calcineurin Inhibitors for Treatment of Steroid-resistant aGVHD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Southern Medical University, China (Other); Peking University People's Hospital (Other); Huazhong University of Science and Technology (Other); Sun Yat-sen University (Other); Academy Military Medical Science, China (Industry)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSC-aGVHD-2014
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Acute Graft-versus-host Disease
Keywords: Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells; CD25 Monoclonal Antibody; Acute Graft-versus-host disease
MeSH Terms: interventions — PC61 monoclonal antibody; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cells (Experimental): MSCs will be given at a median dose of 1×10^6 cells/kg once weekly for 4 dose (as 1 cycle) or until CR. The response should be evaluated at 3 and 4 weeks. If symptoms of aGVHD progress at 3 weeks or the patients have NR at 4 weeks, these patients will switch to other therapy. If patients achieved PR at 4 weeks, another cycle will be given. Besides, CD25 monoclonal antibody (20mg/kg) will be administered at day 1,4,8,15, 21 and calcineurin inhibitors will also be used.
  Interventions: Drug: CD25 monoclonal antibody; Drug: calcineurin inhibitors; Biological: MSCs
- CD25 Mc Ab & calcineurin inhibitors (Experimental): CD25 monoclonal antibody (20mg/kg, day 1,4,8,15,21) will be administered combined with calcineurin inhibitors. The response should be evaluated at 3 and 4 weeks. If symptoms of aGVHD progress at 3 weeks or the patients have NR at 4 weeks, these patients will switch to other therapy. If patients achieved PR at 4 weeks, another cycle will be given.
  Interventions: Drug: CD25 monoclonal antibody; Drug: calcineurin inhibitors

INTERVENTIONS:
Drug: CD25 monoclonal antibody
Drug: calcineurin inhibitors
Biological: MSCs
  Arms: Mesenchymal stem cells

SUMMARY:
The purpose of this study is to compare the efficacy of CD25 monoclonal antibody and calcineurin inhibitors with or without mesenchymal stem cells (MSCs) in treating patients with steroid-resistant acute graft-versus-host disease (aGVHD) after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective therapy for several hematological disorders. Although good progress has been made in the prevention and treatment of side effects associated with transplantation, aGVHDremains a common and life-threatening complication with poor prognosis. Corticosteroids are still acted as the first-line treatments of aGVHD, with a response rate of 50-80. However, those who failed to initial therapy only have 10-30% long-term survival.

Mesenchymal stromal cells (MSCs) are a form of multipotent adult stem cells that can be isolated from many tissues, such as bone marrow (BM), adipose tissue and umbilical cord. Such cells possess the capacity to suppress immunological responses, support hematopoiesis and repair tissues. Clinical applications of human MSCs are evolving rapidly for preventing and treating GVHD. Although the results are still controversy, most prospective and retrospective data suggest that MSCs are effective to aGVHD.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded BM-derived MSCs from third-party donors combined with CD25 monoclonal antibody and calcineurin inhibitors in treating patients with aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* age of 14-65 years
* steroid-resistant aGVHD
* subjects (or their legally acceptable representatives) must have signed an informed consent document

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of treatment for steroid-resistant aGVHD | 1 year
  The responses to aGVHD are according to the literature criteria, including completely response (CR), partial response (PR) and no response (NR), and CR is defined as resolution of all symptoms of aGVHD; PR is defined as a decrease by at least 1 GVHD stage in any 1 organ system without deterioration in others 24. Overall response (OR) includes CR and PR.

SECONDARY OUTCOMES:
Incidence of infections | 1 year
  Infections are mainly focused on cytomegalovirus (CMV) and Epstein-Barr virus ( EBV) infections during study treatments and within one year after study treatments.
Incidence of primary underlying disease relapse | 1 year
Incidence of chronic GVHD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Le Blanc K, Rasmusson I, Sundberg B, Gotherstrom C, Hassan M, Uzunel M, Ringden O. Treatment of severe acute graft-versus-host disease with third party haploidentical mesenchymal stem cells. Lancet. 2004 May 1;363(9419):1439-41. doi: 10.1016/S0140-6736(04)16104-7. PMID 15121408
- [Background] Perez-Simon JA, Lopez-Villar O, Andreu EJ, Rifon J, Muntion S, Diez Campelo M, Sanchez-Guijo FM, Martinez C, Valcarcel D, Canizo CD. Mesenchymal stem cells expanded in vitro with human serum for the treatment of acute and chronic graft-versus-host disease: results of a phase I/II clinical trial. Haematologica. 2011 Jul;96(7):1072-6. doi: 10.3324/haematol.2010.038356. Epub 2011 Mar 10. PMID 21393326
- [Derived] Zhao K, Lin R, Fan Z, Li Z, Chen X, Xuan L, Huang F, Xu N, Wu X, Chen S, Sun J, Zhang X, Weng J, Li Y, Li Y, Lin D, Nie D, Wang S, Xu X, Zhang X, Li Y, Xiang AP, Wang Y, Liu Q. Reduced morbidity and mortality of cGVHD in patients who received treatment with mesenchymal stromal cells for steroid-resistant aGVHD: long-term follow-up of a randomized phase 3 trial. Exp Hematol Oncol. 2025 Jul 9;14(1):95. doi: 10.1186/s40164-025-00687-8. PMID 40635107
- [Derived] Zhao K, Lin R, Fan Z, Chen X, Wang Y, Huang F, Xu N, Zhang X, Zhang X, Xuan L, Wang S, Lin D, Deng L, Nie D, Weng J, Li Y, Zhang X, Li Y, Xiang AP, Liu Q. Mesenchymal stromal cells plus basiliximab, calcineurin inhibitor as treatment of steroid-resistant acute graft-versus-host disease: a multicenter, randomized, phase 3, open-label trial. J Hematol Oncol. 2022 Mar 7;15(1):22. doi: 10.1186/s13045-022-01240-4. PMID 35255929